CLINICAL TRIAL: NCT06485518
Title: Integration of the 5G-based Remote Healthcare System in Critical Care: A Comprehensive Report With Multiple Satellite Sites
Brief Title: Integration of the 5G-based Remote Healthcare System in Critical Care
Acronym: IT5GRHSCI
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yucai Hong, PI, Sir Run Run Shaw Hospital
Other Study IDs: ky20220304-31; 2023YFC3603100 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Emergency Medicine; Telemedicine; Augmented Reality
Keywords: Teleconference; Mentoring; Augmented Reality; Emergency; Patient outcome
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5G RHS group: For all patients receiving care through the 5G-based Remote Healthcare System (5G RHS) teleconsultation platform during the specified time period
  Interventions: Behavioral: The 5G RHS group receiving audio-video conferencing and effective data management for decision-making via augmented reality platform RealHealthcare System.

INTERVENTIONS:
Behavioral: The 5G RHS group receiving audio-video conferencing and effective data management for decision-making via augmented reality platform RealHealthcare System. — The 5G RHS group will receive audio-video conferencing and effective data management for decision-making via augmented reality platform. A total of 14 physicians from SRRSH will be participated in the study, offering remote consultations and instant guidance to the physician.

SUMMARY:
The primary objective of this initial report is to address the following questions: Under what circumstances do clinical teams at satellite locations utilize the 5G RHS? Does the implementation of 5G RHS result in significant clinical enhancements? Furthermore, additional analyses will be conducted to assess specific improvements in various use cases (e.g., emergency room, diagnosis, treatment, task guidance, and medical education) and to examine whether factors such as the expertise of central physicians, patient and physician locations, and the timing of calls influence clinical outcomes.

DETAILED DESCRIPTION:
Background: Augmented Reality (AR) has undergone rapid development in recent years, gaining prominence in healthcare, especially when coupled with 5G internet technology. This study delves into the integration of 5G Augmented Reality in emergency medicine, with a focus on its impact on clinical outcomes.

Methods: This study will utilize the 5G-based Remote Healthcare System (5G RHS) to connect four satellite Emergency Room (ER) teams with central experts to assess its effectiveness in critical cases. Data will be collected from July 2022 to June 2023 to address key research questions, including the circumstances prompting the use of 5G RHS, the extent of clinical improvement achieved, and the influence of central physician expertise, patient and physician locations, and calling time on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age range (≥18 years old).
* 2) Patients with acute chest pain, stroke and trauma were diagnosed in the departments of emergency medicine of the relevant medical community, Branches of Run Run Shaw Hospital, Zhejiang University School of Medicine.
* 3) Voluntarily participate in the study and sign the informed consent; If the subject does not have the ability to understand or sign the informed consent, his/her guardian will represent him/her in the informed process and agree to participate in the study; If illiterate, his/her will need a witness to witness the knowledge process and his/her will decide to participate in the study.

Exclusion Criteria:

* 1) Incomplete clinical data.
* 2) Minors.
* 3) Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, patients with acute chest pain, stroke and trauma will be enrolled in the departments of emergency medicine in the relevant medical community, Branches of Run Run Shaw Hospital, Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
critical conditions | from July 2022 to June 2023
  For all patients receiving care through the 5G RHS platform during the specified time period, we gathered clinical data from electronic health records (EHRs). This data encompasses information related to critical conditions.
background situation | from July 2022 to June 2023
  For all patients receiving care through the 5G RHS platform during the specified time period, we will gather clinical data from electronic health records (EHRs). This data encompasses information related to the emergency situation,
reasons for consultation | from July 2022 to June 2023
  For all patients receiving care through the 5G RHS platform during the specified time period, we will gather clinical data from electronic health records (EHRs). This data encompasses information related to reasons for seeking remote consultation (including complex challenges, new medical scenarios, and educational interactions).
treatment outcomes | from July 2022 to June 2023
  For all patients receiving care through the 5G RHS platform during the specified time period, we will gather clinical data from electronic health records (EHRs). This data encompasses information related to treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yecheng Jin, M.D, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
1. The data are not publicly available due to their containing information that could compromise the privacy of research participants.
  2. Data cannot be shared openly but are available on request from authors for some reasonable conditions.